CLINICAL TRIAL: NCT04757922
Title: Stop Ovarian Cancer Young; Effect of the Opportunistic Salpingectomy on Age of Menopause
Acronym: STOPOVCAyoung
Status: Enrolling by invitation | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-6885
Record Dates: First submitted 2021-02-05; First posted 2021-02-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Salpingectomy; Tubal Ligation; Menopause
Keywords: Salpingectomy; Sterilization; Tubal ligation; Opportunistic salpingectomy; Menopausal age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: bilateral salpingectomy: Premenopausal women between 30 and 45 years of age, who will undergo sterilization through Opportunistic Salpingectomy will be asked to participate in the STOPOVCAyoung study.
  Interventions: Procedure: Opportunistic salpingectomy / bilateral salpingectomy
- Control: tubal ligation or no sterilization: The control group will consists of women who chose for sterilization by clips/tubal ligation supplemented by friend/acquaintances, around the same age, who are not planning to undergo sterilization.

INTERVENTIONS:
Procedure: Opportunistic salpingectomy / bilateral salpingectomy — An opportunistic salpingectomy refers to removal of the salpinges without the ovaries during (laparoscopic) interventions for benign (gynaecological) disease to reduce the number of ovarian cancer cases. Therefore, a so-called opportunistic salpingectomy is a method of female sterilization.
  Groups: Intervention: bilateral salpingectomy

SUMMARY:
The aim of this study is to evaluate the long-term safety of on the onset of menopause.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the long-term safety of on the onset of menopause. To investigate the effect of Opportunistic Salpingectomy on the age of menopause, we will compare age of menopause in women who underwent sterilization through opportunistic salpingectomy with a control group consisting of women who underwent sterilization by tubal ligation or who had no sterilization.

ELIGIBILITY:
Inclusion Criteria:

Intervention group

* Undergoing an Opportunistic Salpingectomy as sterilization method
* Premenopausal status at enrolment
* Age between 30 and 45 years
* Will have residual ovarian tissue after surgery
* Able to understand the written or spoken Dutch language
* Gives consent for participating in surveys

Control group

* Premenopausal status at enrolment
* Either sterilization by tubal ligation or no sterilization at all
* Age between 35 and 45 years
* Able to understand the written or spoken Dutch language
* Gives consent for participating in surveys

Exclusion Criteria:

* Postmenopausal status at enrolment
* Under the age of 35 or above 45
* Previous salpingectomy of oophorectomy
* Previous hysterectomy
* Women with abnormal karyotype (such as Turner Syndrome and Fragile X syndrome)
* Underwent chemotherapy or radiation
* Unable to understand the written or spoken Dutch language

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who underwent sterilization (bilateral salpingectomy / tubal ligation) supplemented by friend/acquaintances, around the same age, who are not planning to undergo sterilization.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Menopausal age | At end of follow-up (follow up ends at age of menopause with a maximum follow-up time of 15 years)
  The age of reaching natural menopause (e.g. last menstruation > 1 year ago )

SECONDARY OUTCOMES:
Decision regret | 1 year post surgery and at age of menopause
  The decision regret regarding their choice of sterilization method.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen MJ Piek, MD, PhD, Principal Investigator — Catharina Ziekenhuis; Joanne A de Hullu, MD, PhD, Principal Investigator — University Medical Center Nijmegen
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piek JM, van Diest PJ, Zweemer RP, Jansen JW, Poort-Keesom RJ, Menko FH, Gille JJ, Jongsma AP, Pals G, Kenemans P, Verheijen RH. Dysplastic changes in prophylactically removed Fallopian tubes of women predisposed to developing ovarian cancer. J Pathol. 2001 Nov;195(4):451-6. doi: 10.1002/path.1000. PMID 11745677
- [Background] Reade CJ, McVey RM, Tone AA, Finlayson SJ, McAlpine JN, Fung-Kee-Fung M, Ferguson SE. The fallopian tube as the origin of high grade serous ovarian cancer: review of a paradigm shift. J Obstet Gynaecol Can. 2014 Feb;36(2):133-140. doi: 10.1016/S1701-2163(15)30659-9. PMID 24518912
- [Background] Falconer H, Yin L, Gronberg H, Altman D. Ovarian cancer risk after salpingectomy: a nationwide population-based study. J Natl Cancer Inst. 2015 Jan 27;107(2):dju410. doi: 10.1093/jnci/dju410. Print 2015 Feb. PMID 25628372
- [Background] van Lieshout LAM, Steenbeek MP, De Hullu JA, Vos MC, Houterman S, Wilkinson J, Piek JM. Hysterectomy with opportunistic salpingectomy versus hysterectomy alone. Cochrane Database Syst Rev. 2019 Aug 28;8(8):CD012858. doi: 10.1002/14651858.CD012858.pub2. PMID 31456223
- [Background] Hanley GE, Kwon JS, Finlayson SJ, Huntsman DG, Miller D, McAlpine JN. Extending the safety evidence for opportunistic salpingectomy in prevention of ovarian cancer: a cohort study from British Columbia, Canada. Am J Obstet Gynecol. 2018 Aug;219(2):172.e1-172.e8. doi: 10.1016/j.ajog.2018.05.019. Epub 2018 May 28. PMID 29852159
- [Background] McAlpine JN, Tone AA, Hanley GE. Opportunistic Salpingectomy: We Chose to Act, Not Wait. J Obstet Gynaecol Can. 2016 May;38(5):425-7. doi: 10.1016/j.jogc.2016.04.084. Epub 2016 May 6. No abstract available. PMID 27261215
- [Derived] Gelderblom ME, IntHout J, Hermens RPMG, Coppus SFPJ, Ebisch I, van Ginkel AA, van de Laar R, de Lange N, Maassen M, Pijlman B, Smedts HPM, Vos MC, Beerendonk CCM, de Hullu JA, Piek JMJ. STop OVarian CAncer (STOPOVCA) young: Protocol for a multicenter follow-up study to determine the long-term effects of opportunistic salpingectomy on age at menopause. Maturitas. 2022 May;159:62-68. doi: 10.1016/j.maturitas.2022.01.006. Epub 2022 Jan 15. PMID 35337614